CLINICAL TRIAL: NCT04460313
Title: Observatory of Nasopharyngeal Carriage of Streptococcus Pneumoniae (Sp) in Infants With Acute Otitis and in Healthy Child - Ancillary Study for Detection of E Coli ESBL Carriers
Brief Title: Nasopharyngeal Carriage of S. Pneumoniae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACT0806
Record Dates: First submitted 2020-06-19; First posted 2020-07-07 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Nasopharyngeal Carriage; Children, Only; Antibiotic Resistant Strain
Keywords: Pneumococcal conjugate vaccine; Streptococcus pneumoniae; Carriage

STUDY DESIGN:
Intervention Model Description: multicenter nationwide prospective cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prospective cohort (Other): Nasopharyngeal sample for each enrolled children
  Interventions: Other: nasopharyngeal sample
- ESBL cohort (Other): Stool or anorectal swab samples for a subgroup of children
  Interventions: Other: nasopharyngeal sample; Other: Stools collection or anorectal swab samples

INTERVENTIONS:
Other: nasopharyngeal sample — Nasopharyngeal swabs from children with acute otitis media aged 6 to 24 months. The swabs were analyzed by the French National Reference Centre for Pneumococci.
Other: Stools collection or anorectal swab samples — For a subgroup of children stools samples or anorectal swab samples were collected for assessment of E. coli (ESBL) resistance
  Arms: ESBL cohort

SUMMARY:
This nasopharyngeal (NP) carriage surveillance study was requested by the European Agency for the Evaluation of Medicinal Products as a post-licensing commitment to determine whether the use of the pneumococcal conjugate vaccines (PCVs) including 7 then 13 valents (introduced in 2001 and 2010, respectively) caused a shift in the distribution of Streptococcus pneumoniae serotypes in children with acute otitis media and modified the resistance of this bacterial species to antibiotics.

DETAILED DESCRIPTION:
Since September 2001, 121 pediatricians who are part of a research and teaching network (ACTIV) throughout France participated at this prospective study. From October to June of each subsequent year, children of both sexes suffering from suppurative acute otitis media (AOM) with fever and/or otalgia (in order to increase the probability of pneumococcal AOM), aged 6 to 24 months, were enrolled.

And a second group of healthy children aged 6 months to 15 years were also enrolled for the main study.

For ancillary study a subgroup of children were enrolled for assessment of E. coli (ESBL) resistance.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* suffering from suppurative AOM
* age: 6 months to 24 months for AOM
* age: 6 months to 15 years for healthy children
* informed consent from parents or guardians

Exclusion Criteria:

* Children with antibiotic treatment within 7 days before enrolment,
* severe underlying disease,
* inclusion in the study during the previous 12 months

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23560 (Estimated)
Dates: Start 2001-09-11 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
S. Pneumoniae colonisation to detect emerging serotypes | at inclusion
  The percentage of children colonised by non vaccine serotypes -

SECONDARY OUTCOMES:
Detect the emergence of resistance S. pneumoniae | at inclusion
  Percentage of penicillin resistant S. pneumoniae
Evaluation of the rhinopharyngeal carriage of other bacteria | at inclusion
  Haemophilus influenzae, Moraxella Catarrhalis, and Staphylococcus aureus in AOM group and healthy children.
Detect the emergence of new serotypes | at inclusion
  > 10 Percent of isolated Sp, 5 percent of carrier children
For the ancillary study, the resistance of E. coli (ESBL) will be evaluated. | at inclusion
  Assessment of E. coli (ESBL) resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cohen, MD, Principal Investigator — Association Clinique Thérapeutique Infantile du val de Marne
Locations (1):
- ACTIV, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ouldali N, Cohen R, Levy C, Gelbert-Baudino N, Seror E, Corrard F, Vie Le Sage F, Michot AS, Romain O, Bechet S, Bonacorsi S, Angoulvant F, Varon E. Pneumococcal susceptibility to antibiotics in carriage: a 17 year time series analysis of the adaptive evolution of non-vaccine emerging serotypes to a new selective pressure environment. J Antimicrob Chemother. 2019 Oct 1;74(10):3077-3086. doi: 10.1093/jac/dkz281. PMID 31280295
- [Result] Rybak A, Levy C, Bonacorsi S, Bechet S, Vie le Sage F, Elbez A, Varon E, Cohen R. Antibiotic Resistance of Potential Otopathogens Isolated From Nasopharyngeal Flora of Children With Acute Otitis Media Before, During and After Pneumococcal Conjugate Vaccines Implementation. Pediatr Infect Dis J. 2018 Mar;37(3):e72-e78. doi: 10.1097/INF.0000000000001862. PMID 29227464
- [Result] Birgy A, Bidet P, Levy C, Sobral E, Cohen R, Bonacorsi S. CTX-M-27-Producing Escherichia coli of Sequence Type 131 and Clade C1-M27, France. Emerg Infect Dis. 2017 May;23(5):885. doi: 10.3201/eid2305.161865. No abstract available. PMID 28418829
- [Result] Cohen R, Varon E, Doit C, Schlemmer C, Romain O, Thollot F, Bechet S, Bonacorsi S, Levy C. A 13-year survey of pneumococcal nasopharyngeal carriage in children with acute otitis media following PCV7 and PCV13 implementation. Vaccine. 2015 Sep 22;33(39):5118-26. doi: 10.1016/j.vaccine.2015.08.010. Epub 2015 Aug 11. PMID 26271823
- [Result] Cohen R, Levy C, Bonnet E, Thollot F, Boucherat M, Fritzell B, Derkx V, Bingen E, Varon E. Risk factors for serotype 19A carriage after introduction of 7-valent pneumococcal vaccination. BMC Infect Dis. 2011 Apr 18;11:95. doi: 10.1186/1471-2334-11-95. PMID 21501471
- [Result] Cohen R, Bingen E, Levy C, Thollot F, Boucherat M, Derkx V, Varon E. Nasopharyngeal flora in children with acute otitis media before and after implementation of 7 valent pneumococcal conjugate vaccine in France. BMC Infect Dis. 2012 Mar 7;12:52. doi: 10.1186/1471-2334-12-52. PMID 22397629
- [Result] Levy C, Vie le Sage F, Varon E, Chalumeau M, Grimprel E, Cohen R. Pediatric Ambulatory and Hospital Networks for Surveillance and Clinical Epidemiology of Community-Acquired Infections. J Pediatr. 2018 Mar;194:269-270.e2. doi: 10.1016/j.jpeds.2017.11.050. Epub 2018 Feb 22. No abstract available. PMID 29637893
- [Result] Vermee Q, Cohen R, Hays C, Varon E, Bonacorsi S, Bechet S, Thollot F, Corrard F, Poyart C, Levy C, Raymond J. Biofilm production by Haemophilus influenzae and Streptococcus pneumoniae isolated from the nasopharynx of children with acute otitis media. BMC Infect Dis. 2019 Jan 11;19(1):44. doi: 10.1186/s12879-018-3657-9. PMID 30634919
- [Result] Birgy A, Madhi F, Jung C, Levy C, Cointe A, Bidet P, Hobson CA, Bechet S, Sobral E, Vuthien H, Ferroni A, Aberrane S, Cuzon G, Beraud L, Gajdos V, Launay E, Pinquier D, Haas H, Desmarest M, Dommergues MA, Cohen R, Bonacorsi S; Group of the National Observatory of Urinary tract Infection due to ESBL-producing Enterobacteriaceae in children. Diversity and trends in population structure of ESBL-producing Enterobacteriaceae in febrile urinary tract infections in children in France from 2014 to 2017. J Antimicrob Chemother. 2020 Jan 1;75(1):96-105. doi: 10.1093/jac/dkz423. PMID 31617912
- [Result] Mizrahi A, Cohen R, Varon E, Bonacorsi S, Bechet S, Poyart C, Levy C, Raymond J. Non typable-Haemophilus influenzae biofilm formation and acute otitis media. BMC Infect Dis. 2014 Jul 19;14:400. doi: 10.1186/1471-2334-14-400. PMID 25037572
- [Result] Birgy A, Levy C, Bidet P, Thollot F, Derkx V, Bechet S, Mariani-Kurkdjian P, Cohen R, Bonacorsi S. ESBL-producing Escherichia coli ST131 versus non-ST131: evolution and risk factors of carriage among French children in the community between 2010 and 2015. J Antimicrob Chemother. 2016 Oct;71(10):2949-56. doi: 10.1093/jac/dkw219. Epub 2016 Jun 20. PMID 27330068
- [Result] Hau I, Levy C, Caeymaex L, Cohen R. Impact of pneumococcal conjugate vaccines on microbial epidemiology and clinical outcomes of acute otitis media. Paediatr Drugs. 2014 Feb;16(1):1-12. doi: 10.1007/s40272-013-0044-2. PMID 23963858
- [Result] Birgy A, Cohen R, Levy C, Bidet P, Courroux C, Benani M, Thollot F, Bingen E. Community faecal carriage of extended-spectrum beta-lactamase-producing Enterobacteriaceae in French children. BMC Infect Dis. 2012 Nov 21;12:315. doi: 10.1186/1471-2334-12-315. PMID 23171127
- [Result] Caeymaex L, Varon E, Levy C, Bechet S, Derkx V, Desvignes V, Doit C, Cohen R. Characteristics and outcomes of acute otitis media in children carrying streptococcus pneumoniae or haemophilus influenzae in their nasopharynx as a single otopathogen after introduction of the heptavalent pneumococcal conjugate vaccine. Pediatr Infect Dis J. 2014 May;33(5):533-6. doi: 10.1097/INF.0000000000000213. PMID 24263220
- [Result] Cohen R, Levy C, Bingen E, Koskas M, Nave I, Varon E. Impact of 13-valent pneumococcal conjugate vaccine on pneumococcal nasopharyngeal carriage in children with acute otitis media. Pediatr Infect Dis J. 2012 Mar;31(3):297-301. doi: 10.1097/INF.0b013e318247ef84. PMID 22330166
- [Result] Cohen R, Levy C, Bingen E, Bechet S, Derkx V, Werner A, Koskas M, Varon E. [Nasopharyngeal carriage of children 6 to 60 months during the implementation of the 13-valent pneumococcal conjugate vaccine]. Arch Pediatr. 2012 Oct;19(10):1132-9. doi: 10.1016/j.arcped.2012.07.013. Epub 2012 Aug 24. French. PMID 22925540
- [Result] Cohen R, Levy C, Thollot F, de La Rocque F, Koskas M, Bonnet E, Fritzell B, Varon E. Pneumococcal conjugate vaccine does not influence Staphylococcus aureus carriage in young children with acute otitis media. Clin Infect Dis. 2007 Dec 15;45(12):1583-7. doi: 10.1086/523734. PMID 18190319
- [Result] Cohen R, Levy C, de La Rocque F, Gelbert N, Wollner A, Fritzell B, Bonnet E, Tetelboum R, Varon E. Impact of pneumococcal conjugate vaccine and of reduction of antibiotic use on nasopharyngeal carriage of nonsusceptible pneumococci in children with acute otitis media. Pediatr Infect Dis J. 2006 Nov;25(11):1001-7. doi: 10.1097/01.inf.0000243163.85163.a8. PMID 17072121
- See also: ACTIV publications — https://www.activ-france.com/fr/publications